CLINICAL TRIAL: NCT06203769
Title: Reduction of Antibiotherapy Duration for Infections on Implantable Extra Cardiac Devices Leads: a Randomized Controlled Multicenter Non-inferiority Trial
Brief Title: Reduction of Antibiotherapy Duration for Infections on Implantable Extra Cardiac Devices Leads
Acronym: RAID
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP220013
Record Dates: First submitted 2023-11-29; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Cardiac Devices Infection
Keywords: Infections; Antibiotherapy; Implantable extra cardiac devices; Non-inferiority; Randomized
MeSH Terms: conditions — Infections | interventions — Anti-Infective Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 14-day antibiotic therapy after removal of infected material
  Interventions: Drug: 14-day antibiotic therapy
- control group (Active Comparator): 28-day antibiotic therapy after removal of infected material
  Interventions: Drug: 28-day antibiotic therapy

INTERVENTIONS:
Drug: 14-day antibiotic therapy — The studied intervention will be 14-day antibiotic therapy after removal of infected material
  Other Names: Experimental arm
  Arms: Experimental group
Drug: 28-day antibiotic therapy — The comparator arm will be 28-day antibiotic therapy after removal of infected material
  Other Names: Control arm
  Arms: control group

SUMMARY:
The design is an Open-label randomized controlled multicenter non-inferiority trial with blinded assessor which compares 2 antibiotic strategy: 14-day antibiotic therapy after removal of infected material (experimental group) versus 28-day antibiotic therapy after removal of infected material (control group).

Randomization will be centralized, individual 1:1, stratified on center and age (<75 versus >=75 years). Analysis will be reported following CONSORT guidelines for pharmacological trials.

Main analysis will be conducted according to per protocol and intent-to-treat principles. Subgroup analysis will be conducted according to age, classes of antibiotics at baseline and according to resistance testing and baseline renal clearance.

DETAILED DESCRIPTION:
Infections of cardiac implantable electronic devices (CIED) are one of the most frequent complication after implantation of these devices, with an incidence rate estimated at 4.82 / 1000 in Denmark, mainly in the first year post implantation. An american study found that the incidence of CIED infection in the USA increased from 1.53% in 2004 to 2.41% in 2008 and a National Inpatient Sample database study showed an increase from 1.45% to 3.41% (P<0.001) from 2000 through 2012. These figures are constantly increasing and concern mostly older people.

Although the mortality seems to be low compared to those of valvular infection , evaluated at 4% for nonstaphylococcal infection and up to 9% for Staphylococcus aureus related infections, those infections are responsible of numerous morbidities such as iterative hospitalizations, decompensations of other comorbidities and autonomy loss, especially, for older people

Clinical presentations of CIED infections are varied and include generator pocket infections, native or prosthetic CIED-associated valvular endocarditis (CIED-IE) with echocardiographic evidence of valve involvement, and CIED lead infections (CIED-LI) with evidence of lead infection without valve involvement.

In CIED infections, removal of the device is the cornerstone of treatment and is usually required to enable cure in association with antimicrobial therapy for a few weeks. However, although antimicrobial therapy duration after removal of the device are relatively well defined for generator pocket infections (10 - 14 days for the remaining skin and soft tissue infection) and CIED-IE (4 - 6 weeks), the optimal duration of antibiotic treatment in CIED-LI has yet to be determined.

Several series amalgamate generator pocket infection, CIED-IE and CIED-LI descript duration of therapy and are therefore unhelpful in deciding on the optimum duration of antimicrobials.

Guidelines for management of CIED infections recommend different durations of antibiotic treatment, particularly for CIED-LI, which can result in considerable inappropriate antimicrobial exposure in a vulnerable patient population.

In light of the emergence of bacterial resistance and in order to limit the drug toxicities of antibiotics, it is crucial to offer patients the shortest possible duration of treatment, without losing efficiency.

Infections of cardiac implantable electronic devices (CIED) are one of the most frequent complication after implantation of these devices, with an incidence rate estimated at 4.82 / 1000 in Denmark, mainly in the first year post implantation(1). An american study found that the incidence of CIED infection in the USA increased from 1.53% in 2004 to 2.41% in 2008 and a National Inpatient Sample database study showed an increase from 1.45% to 3.41% (P<0.001) from 2000 through 2012. These figures are constantly increasing and concern mostly older people.

Although the mortality seems to be low compared to those of valvular infection , evaluated at 4% for nonstaphylococcal infection and up to 9% for Staphylococcus aureus related infections (4), those infections are responsible of numerous morbidities such as iterative hospitalizations, decompensations of other comorbidities and autonomy loss, especially, for older people

Clinical presentations of CIED infections are varied and include generator pocket infections, native or prosthetic CIED-associated valvular endocarditis (CIED-IE) with echocardiographic evidence of valve involvement, and CIED lead infections (CIED-LI) with evidence of lead infection without valve involvement.

In CIED infections, removal of the device is the cornerstone of treatment and is usually required to enable cure in association with antimicrobial therapy for a few weeks. However, although antimicrobial therapy duration after removal of the device are relatively well defined for generator pocket infections (10 - 14 days for the remaining skin and soft tissue infection) and CIED-IE (4 - 6 weeks) (5), the optimal duration of antibiotic treatment in CIED-LI has yet to be determined.

Several series amalgamate generator pocket infection, CIED-IE and CIED-LI descript duration of therapy and are therefore unhelpful in deciding on the optimum duration of antimicrobials .

Guidelines for management of CIED infections recommend different durations of antibiotic treatment, particularly for CIED-LI, which can result in considerable inappropriate antimicrobial exposure in a vulnerable patient population.

In light of the emergence of bacterial resistance and in order to limit the drug toxicities of antibiotics, it is crucial to offer patients the shortest possible duration of treatment, without losing efficiency.

To this regard, renal failure is one of the most frequent adverse effect during antibiotic treatment, especially in older patients with polymedication and comorbidities, and is responsible indirectly of increasing mortality.

Furthermore, shortening antibiotic therapy would allow to decrease the number of allergy events and Clostridium difficile colitis.

In the most recent European recommendations , if the TEE performed after device removal shows no signs of valve vegetation (i.e. isolated lead vegetation), the follow-up blood cultures are negative, the clinical improvement is good and there are no pulmonary abscesses, treatment duration for 2 weeks post-device extraction can be sufficient but total treatment duration should not be shorter than 4 weeks.

Older U.S guidelines recommend at least 2 weeks of parenteral therapy after extraction of an infected device for patients with bloodstream infection. Patients with sustained (>24 hours) positive blood cultures despite CIED removal and appropriate antimicrobial therapy should receive parenteral therapy for at least 4 weeks, even if TEE is negative for valvular vegetations.

In the British recommendations short course therapy (2 weeks) could be considered if tricuspid valve is structurally normal, no ghost lesions present after system removal on control TEE and rapid clinical response to device removal.

Finally, no clinical trial data are available to define the optimal duration of antimicrobial therapy for CIED-LI and all recommendations are based on retrospective studies and expert opinion. U.S guidelines are mainly based on one retrospective, non-randomized, monocenter cohort study leading to possible confusion and indication bias. However, this study, which is to our knowledge the only one on this topic, 189 patients were included from 1991 to 2003 and presented either a generator pocket infections, a CIED-IE, or a CIED-LI without valvular infection. All results were "pooled" together when describing duration of therapy and are therefore unhelpful in deciding on the optimum duration of antimicrobials. Besides, english recommendations are based on expert opinions, themselves based on case series and pharmacological considerations .

Our hypothesis is therefore that in CIED-LI, 14 days of antimicrobial therapy after device extraction is sufficient regardless of the duration of previous antibiotic therapy if the bacteremia is controlled and if there are (i) no distant infectious foci (abscess), no valvular lesions

Therefore the benefit-risk balance of a shortening of antibiotic therapy for CIED infections needs to be assessed with a high-level of evidence.

This study is endorsed by AEPEI

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of CIED leads infections, defined by:

  1. Symptoms/signs of systemic infection AND positive blood cultures fulfilled the major Duke microbiological criteria AND echocardiography consistent with vegetation(s) attached to lead(s) AND/OR [18F]FDG PET/CT or radiolabelled WBC SPECT/CT detection of abnormal activity along leads OR
  2. Symptoms/signs of systemic infection AND NO, signs of generator pocket infection, AND culture, histology or molecular evidence of infection on explanted lead.
* Complete removal of the infected CIED
* Signed informed consent
* French National Health Assurance

Exclusion Criteria:

* Current involvement of native or prosthetic heart valve
* Distant infectious foci (such as haematogenous vertebral osteomyelitis, pulmonary abscess…) justifying a prolonged duration of therapy.
* Positive blood culture > 24 hours after cultures despite CIED removal
* CIED infection with Mycobacteria or Fungi
* Women who are pregnant or nursing
* Females of childbearing potential without effective method of birth control
* Patients who are under tutorship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Mortality, | at 3 months after randomization,
  Mortality linked to infection during or after antibiotic therapy
Rate of relapse of infection | at 3 months after randomization
  Rate of relapse of infection defined by diagnostic of endocarditis or CIED infection with the same bacteria
Rate of relapse of infection | at 6 months after randomization
  Number of patient whith relapse of infection defined by diagnostic of endocarditis or CIED infection with the same bacteria
Rate of a distant infections | at 3 months after randomization
  Rate of a distant infectious foci with the same bacteria
Rate of a distant infectious | 6 months after randomization
  Rate of diagnostic of a distant infectious foci with the same bacteria

SECONDARY OUTCOMES:
Rate of Acute Renal failure, | at the end of the antibiotherapy period
  rate of Acute Renal failure at the end of the antibiotherapy
Rate of Acute Renal failure, | at 3 months after the end of the antibiotherapy
  Rate of Acute Renal failure at 3 months after the end of the antibiotherapy antibiotherapy
Rate of Acute Renal failure, | at 6 months after the end of the antibiotherapy
  The Rate of Acute Renal failure at 6 months after the end of the antibiotherapy
Rate of Clostridium difficile colitis, | at 3 months after the end of antibiotherapy
  The measurements of the event occuring will be taken at 3 months after the end of the antibiotherapy périod
Rate of Clostridium difficile colitis, | at 6 months after the end of antibiotherapy
  The measurements of the event occuring will be taken at 6 months afte rthe end of the antibiotherapy périod
Rate of allergy grade III or IV | at 3 months after the end of antibiotherapy
  The measurements of the event occuring will be taken at 3 months after the end of the antibiotherapy périod
Rate of allergy grade III or IV | at 6 months after the end of antibiotherapy
  The measurements of the event occuring will be taken at 6 months after the end of the antibiotherapy périod
Percentage of unplanned hospitalization | within 6 months after the end of antibiotherapy
  Percentage of unplanned hospitalization within 6 months after the end of antibiotherapy
Percentage of emergency consultation, | within 6 months after the end of antibiotherapy
  Percentage of emergency consultation within 6 months after the end of antibiotherapy
percentage of adverse events related to antibiotherapy | within 6 months after the end of antibiotherapy
  Percentage of adverse events related to antibiotherapy within 6 months after the end of antibiotherapy

IPD SHARING:
Plan to Share IPD: No